CLINICAL TRIAL: NCT06000800
Title: Timing of Umbilical Cord Clamping in Preterm Neonates: A Randomized Controlled Trial
Brief Title: Timing of Umbilical Cord Clamping in Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Zaghloul, Lecturer of maternal and newborn health nursing, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Cord Clamping
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cord Clamping
Keywords: Umbilical cord clamping; Preterm Neonates; Randomized Controlled Trial

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial was used to fulfill the aim of the study. The randomized control trial (RCT) is a trial in which subjects are randomly assigned to one of two groups: one (the experimental group) receiving the intervention that is being tested, and the other (the comparison group or control group) receiving an alternative treatment
Masking Description: The trial was unblinded; where the participants and researchers were aware of the group a participant belonged to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group (clamping at 30 seconds) (Experimental): Umbilical cord clamping at 30 seconds
  Interventions: Other: Group B
- Group clamping at 60 seconds (Experimental): Umbilical cord clamping at 60 seconds
  Interventions: Other: Group C
- Group clamping at 90 seconds (Experimental): Umbilical cord clamping at 90 seconds
  Interventions: Other: Group D
- Group clamping immediately (Active Comparator): Umbilical cord clamping immediately after birth (5 second)
  Interventions: Other: Group A

INTERVENTIONS:
Other: Group B — Umbilical cord clamping at 30 seconds
  Arms: Group (clamping at 30 seconds)
Other: Group C — Umbilical cord clamping at 60 seconds
  Arms: Group clamping at 60 seconds
Other: Group D — Umbilical cord clamping at 90 seconds
  Arms: Group clamping at 90 seconds
Other: Group A — Umbilical cord clamping immediately after birth (5 second)
  Arms: Group clamping immediately

SUMMARY:
Umbilical cord clamping is an important intervention that routinely done for all neonates afterbirth. yet the optimal timing for this intervention remains controversial

DETAILED DESCRIPTION:
The study was a randomized controlled trial to assess the effect of timing of umbilical cord clamping on preterm neonatal outcome together The study was conducted in Kasr Al Ainy maternity hospital, Cairo university hospitals which provides free obstetrics and gynecology health services including antepartum, intraparturm, postpartum, and neonatal care for both low risk and high-risk pregnant women A total of 80 pregnant women out of 120 meeting the eligibility criteria were randomly pooled using computer-generated random numbers.

The 80 randomly recruited ladies were randomly allocated using sealed envelopes to a group from 4 equal groups (group A, B, C, and D) of 20 ladies each. Umbilical cord clamping was performed immediately after birth (5 second) in group A, at 30 seconds in group B, at 60 seconds in group C, and at 90 seconds in group D.The trial was unblinded; where the participants and researchers were aware of the group a participant belonged to.

After the study protocol was granted the ethical approval from the research ethical committee of Faculty of Nursing, Cairo University, Egypt, a written informed consent was obtained form mothers of preterm neonate who met the inclusion criteria including the aim, procedure, benefits, and nature of the study .The anonymity and confidentiality of information was assured, and the mothers had the right to withdraw from the study at any time during the study without any effect on the care provided to their preterm neonates.

All study subjects were interviewed using a Structured interview questionnaire to obtain full history to assess participants' demographic data such as age, residence, educational level and occupation, past medical and surgical history, and obstetric history such as gravidity, parity, and current pregnancy antenatal care.

Immediately after birth, neonates in all groups are held 20 cm below the incision level.For neonates in group A,umbilical cord was clamped and cut immediately after birth (5 second); while, neonates in group B, umbilical cord were clamped and cut at 30 seconds. For neonates in group C, umbilical cord was clamped and cut at 60 seconds. And finally, neonates in group D, umbilical cord were clamped and cut at 90 seconds. After cord clamping, all neonates were subject to routine immediate care.

Neonatal data recorded included neonatal characteristic such as gestational age,birth weight and gender.Neonatal condition was assessed and documented immediately after birth through applying APGAR score of neonatal life, birth weight was measured immediately after delivery through birth scale. Vital signs (respiration, pulse & temperature) were measured birth.

A pilot study was conducted on 10% of the study subjects. Eight preterm neonates who met the inclusion criteria; the pilot study was carried out to test the clarity of the tool's questions, and time needed to complete the tools. Additionally, to examine the applicability of the study tool, and to identify any difficulties that may arise and need to be handled before data collection. The pilot study revealed that the tools did not require modification. The sample included in the pilot study was excluded from the main study sample.

The collected data will be coded and statistically analyzed to obtain mean and standard deviation for quantitative variables and frequencies (number of cases) and relative frequencies (percentages) for categorical variables. Comparisons between groups will bedone using analysis of variance (ANOVA) with multiple comparisons post hoc test in normally distributed quantitative variables while non-parametric Kruskal-Wallis test and Mann-Whitney test will be used for non-normally distributed quantitative variables . For comparing categorical data, Chi square test will be performed.

ELIGIBILITY:
Inclusion Criteria

* healthy pregnant mothers
* singleton fetuses
* preterm cesarian delivery

Exclusion Criteria:

* asphyxiated neonates
* twins
* mothers with any medical or obstetrical conditions occurring intrapartum such as hemorrhage, or eclampsia.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
neonatal APGAR score | 1st, 5th and 10th minutes of life
  quick test performed at 1 and 5 minutes after birth to determine the physical condition of the newborn. The five categories assessed are heart rate, respiratory effort, muscle tone, reflex irritability, and color ( score from 8-10 means normal) score from 7-4 moderate asphyxia, from 1-3 sever asphyxia
neonatal vital signs | 1st,6th,12th, 24th, and 48th hours
  respiration
neonatal vital signs | 1st,6th,12th, 24th, and 48th hours
  pulse
neonatal vital signs | 1st,6th,12th, 24th, and 48th hours
  temperature
neonatal hemoglobin | 1st,6th,12th, 24th, and 48th hours
  measuring this labs for neonate
neonatal hematocrit | 1st,6th,12th, 24th, and 48th hours
  measuring this labs for neonate
neonatal bilirubin level test | 1st,6th,12th, 24th, and 48th hours
  measuring this labs for neonate

SECONDARY OUTCOMES:
blood glucose | 1st,6th,12th, 24th, and 48th hours
  measuring this labs for neonate
oxygen saturation | 1st,6th,12th, 24th, and 48th hours
  measuring this labs for neonate

CONTACTS AND LOCATIONS:
Overall Officials: Lawahez M. Dwedar, lecturer, Study Chair — faculty of nursing; Fatma Atta, lecturer, Study Chair — faculty of medicine
Locations (1):
- Faculty of nursinf, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the study will be shared online
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 months
Access Criteria: will be published on magazine

REFERENCES:
- [Background] Alzaree F, Elbohoty A, Abdellatif M. Early Versus Delayed Umbilical Cord Clamping on Physiologic Anemia of the Term Newborn Infant. Open Access Maced J Med Sci. 2018 Aug 15;6(8):1399-1404. doi: 10.3889/oamjms.2018.286. eCollection 2018 Aug 20. PMID 30159064
- [Background] American College of Obstetricians and Gynecologists' Committee on Obstetric Practice. Delayed Umbilical Cord Clamping After Birth: ACOG Committee Opinion, Number 814. Obstet Gynecol. 2020 Dec;136(6):e100-e106. doi: 10.1097/AOG.0000000000004167. PMID 33214530
- [Background] Kc A, Rana N, Malqvist M, Jarawka Ranneberg L, Subedi K, Andersson O. Effects of Delayed Umbilical Cord Clamping vs Early Clamping on Anemia in Infants at 8 and 12 Months: A Randomized Clinical Trial. JAMA Pediatr. 2017 Mar 1;171(3):264-270. doi: 10.1001/jamapediatrics.2016.3971. PMID 28114607
- [Background] Bianchi A, Jacobsson B, Mol BW; FIGO Working Group for Preterm Birth. FIGO good practice recommendations on delayed umbilical cord clamping. Int J Gynaecol Obstet. 2021 Oct;155(1):34-36. doi: 10.1002/ijgo.13841. PMID 34520061
- [Background] Brown BE, Shah PS, Afifi JK, Sherlock RL, Adie MA, Monterrosa LA, Crane JM, Ye XY, El-Naggar WI; Canadian Neonatal Network; Canadian Preterm Birth Network Investigators. Delayed cord clamping in small for gestational age preterm infants. Am J Obstet Gynecol. 2022 Feb;226(2):247.e1-247.e10. doi: 10.1016/j.ajog.2021.08.003. Epub 2021 Aug 9. PMID 34384773
- [Background] Chiruvolu A, Mallett LH, Govande VP, Raju VN, Hammonds K, Katheria AC. Variations in umbilical cord clamping practices in the United States: a national survey of neonatologists. J Matern Fetal Neonatal Med. 2022 Oct;35(19):3646-3652. doi: 10.1080/14767058.2020.1836150. Epub 2020 Oct 20. PMID 33081557
- [Background] Deindl P, Diemert A. From structural modalities in perinatal medicine to the frequency of preterm birth. Semin Immunopathol. 2020 Aug;42(4):377-383. doi: 10.1007/s00281-020-00805-0. Epub 2020 Aug 25. PMID 32840641